CLINICAL TRIAL: NCT02228473
Title: Effect of Glycopyrrolate and Atropine as Adjuncts to Reversal of Non-Depolarizing Neuromuscular Blocking Agents on Postoperative Catheter-Related Bladder Discomfort
Brief Title: Effect of Glycopyrrolate and Atropine on Catheter-Related Bladder Discomfort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CRBDGlycoAtr
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-08

CONDITIONS: Catheter Site Discomfort; Complications; Anesthesia; Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Glycopyrrolate; Atropine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glycopyrrolate (Experimental): Glycopyrrolate will be administered as the adjuncts of neuromuscular blocker reversal agent.
  Interventions: Drug: Glycopyrrolate
- Atropine (Active Comparator): Atropine will be administered as the adjuncts of neuromuscular blocker reversal agent.
  Interventions: Drug: Atropine

INTERVENTIONS:
Drug: Glycopyrrolate — Glycopyrrolate will be administered.
  Arms: Glycopyrrolate
Drug: Atropine — Atropine will be administered.
  Arms: Atropine

SUMMARY:
We want to evaluate the efficacy of the glycopyrrolate and atropine for the prevention of catheter-related bladder discomfort.

DETAILED DESCRIPTION:
The mechanism of catheter-related bladder discomfort is thought to be related to the muscarinic receptor. The adjuncts to reversal agents such as glycopyrrolate and atropine are known to block the muscarinic receptor in different ways.

We want to evaluate the efficacy of the glycopyrrolate and atropine for the prevention of catheter-related bladder discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for transurethral bladder excision under general anesthesia
* ASA I-III

Exclusion Criteria:

* Foley catheter less than 18 Fr.
* Patients with obstruction of urinary tract
* Patients with neurogenic bladder
* Patients with severe obesity
* Patients with neurologic disorder
* Patients with chronic pain
* Patients with allergic history to atropine or glycopyrrolate

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-02 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Catheter-related bladder discomfort | 1 hour postoperatively
  Catheter-related bladder discomfort will be measured at 1 hour postoperatively (0:none, 1:mild, 2:moderate, 3:severe).

SECONDARY OUTCOMES:
Catheter-related bladder discomfort | 0, 6 and 24 hour postoperatively
  Catheter-related bladder discomfort will be measured at 1 hour postoperatively (0:none, 1:mild, 2:moderate, 3:severe).
Hemodynamic parameters | 0, 1, 5, 10 minute postoperatively
  Mean blood pressure and heart rate will be measured at 0, 1, 5, 10 minute postoperatively. Measurement at 10 minute means Mean blood pressure and heart rate at the admission of post-anesthetic care unit.
Nausea | 0, 1, 6 and 24 hour postoperatively
  Nausea will be measured at 0, 1, 6 and 24 hour postoperatively.
Vomiting | 0, 1, 6 and 24 hour postoperatively
  Vomiting will be measured at 0, 1, 6 and 24 hour postoperatively.
Dry mouth | 0, 1, 6 and 24 hour postoperatively
  Dry mouth will be measured at 0, 1, 6 and 24 hour postoperatively.
Flushing | 0, 1, 6 and 24 hour postoperatively
  Flushing will be measured at 0, 1, 6 and 24 hour postoperatively.
Blurred vision | 0, 1, 6 and 24 hour postoperatively
  Blurred vision will be measured at 0, 1, 6 and 24 hour postoperatively.
Dizziness | 0, 1, 6 and 24 hour postoperatively
  Dizziness will be measured at 0, 1, 6 and 24 hour postoperatively.
Analgesics | 0, 1, 6 and 24 hour postoperatively
  The amount of analgesics will be measured at 0, 1, 6 and 24 hour postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Pyoung Park, PhD, Principal Investigator — Seoul National University of Hospital
Locations (1):
- Seoul National University of Hospital, Seoul, Korea, Republic of, South Korea

REFERENCES:
- [Derived] Kim HC, Lim SM, Seo H, Park HP. Effect of glycopyrrolate versus atropine coadministered with neostigmine for reversal of rocuronium on postoperative catheter-related bladder discomfort in patients undergoing transurethral resection of bladder tumor: a prospective randomized study. J Anesth. 2015 Dec;29(6):831-5. doi: 10.1007/s00540-015-2064-2. Epub 2015 Aug 9. PMID 26254585